CLINICAL TRIAL: NCT04621032
Title: Obstructive Sleep Apnea Destabilizes Myocardial Repolarization Homogeneity
Status: Completed | Type: Observational
Sponsor: Nowodworskie Centrum Medyczne (Other)
Collaborators: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Aleksandra Jarecka-Dobroń, clinical doctor, PhD, Nowodworskie Centrum Medyczne
Other Study IDs: 1
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Obstructive Sleep Apnea; Heart Rhythm Disorder; Obesity, Abdominal
Keywords: Obstructive Sleep Apnea; QT interval; QTV; QTc; repolarisation homogeneity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity, Abdominal | interventions — Electrocardiography, Ambulatory; Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSA +: Patients with visceral obesity and newly diagnosed Obstructive Sleep Apnea (during the study)
  Interventions: Diagnostic Test: Polygraphy monitoring; Diagnostic Test: laboratory tests
- OSA -: Patients with visceral obesity in whom Obstructive Sleep Apnea diagnosis have been excluded (during the study)
  Interventions: Diagnostic Test: Polygraphy monitoring; Diagnostic Test: laboratory tests

INTERVENTIONS:
Diagnostic Test: Polygraphy monitoring — All patients with visceral obesity have been tested for Obstructive Sleep Apnea and heart rhythm disorders by usage of polygraphy and Holter-ECG monitoring.
  Other Names: Holter ECG monitoring
Diagnostic Test: laboratory tests — Blood samples for sodium, potassium, calcium, magnesium concentration and fasting glyceamia assessment hae been taken from all patients with visceral obesity.

SUMMARY:
Literature shows that patients with obesity and Obstructive Sleep Apnea (OSA), both occurring independently, are more likely to develop cardiovascular diseases and sudden cardiac death (SCD). Assuming that ventricular depolarization is more stable than repolarization then QT interval parameters may be used for heart muscle repolarization assessment for those groups of patients.

There were 121 patients included in the study, both - women and men, aging from 35-65 with visceral obesity. Only healthy patients were included - the ones who were not treated for any chronic disease, taking QT elongating drugs, or were not treated with Continuous Positive Airway Pressure (CPAP) therapy at that time.

DETAILED DESCRIPTION:
The current study was a prospective, observational clinical trial performed between September 2016 and August 2019 at a single-center institution specializing in treatment of patients with obstructive sleep apnea. The inclusion criteria were as follows: (1) gender: female or male, (2) age 35-65 years old, (3) visceral obesity, (4) lack of acute or chronic diseases that may have an influence on rhythm or conduction disorders, (5) not undergoing Continuous Positive Airway Pressure therapy (CPAP) or taking drugs that have or may have an influence on QT interval duration [according to Credible Meds list (Woosley et al, 2019)], (6) not consuming grapefruits or grapefruit juice for at least 2 weeks before Holter-ECG examination. Patients, who met all inclusion criteria, underwent subject and physical examination, an over-night Holter-ECG, polygraphy and laboratory biochemical tests (sodium, potassium, calcium, magnesium concentration and fasting glyceamia.

Enrolled patients were asked questions about general frame of mind, daytime and nighttime symptoms that may suggest OSA [according to Epworth Sleepiness Scale (https://epworthsleepinessscale.com/about-the-ess/ access date 08 May 2020)]. All patients were fully physically examined. Neck and waist circumference were measured according to STEPwise Approach to Surveillance (STEPS) by WHO (https://www.who.int/ncds/surveillance/steps/en/. [access date 23 April.2019]. Upon subject examination (snoring and choking feeling during the sleep) a corrected neck circumference was calculated.

Polygraphy was conducted using MED Recorder device by Infoscan company according to AASM guidelines (American Academy of Sleep Medicine, International classification of sleep disorders, 2016). The device registered blood saturation, heart rate, airflow, chest and abdomen movements, body position, snoring and single lead ECG. OSA was diagnosed according to AASM definition (American Academy of Sleep Medicine, Sleep-related breathing disorders in adults, 1999): in every patient with Respiratory Disturbance Index (RDI) ≥ 5/hour and with concomitant OSA sings (Epworth Sleepiness Scale ≥ 11 pts) or with RDI ≥ 15/hour. The minimum time of analyzed data without artifacts had to last at least 6 h.

A Holter-ECG examination was conducted using DMS 300-3A device by Oxford company suitable for Cardioscan 10 system. Registration was made simultaneously with polygraphy, during the night. Chosen QT interval assessment parameters were evaluated upon partially automatically analyzed fragments of ECG records. Only nighttime ECG records were analyzed due to maximum comparability (similar patient's physical activity and minimized, because of limited body movements, artifacts). Moreover, the study aimed to assess a heart's activity simultaneous to sleep breathing disorders. Only ECG strips with constant heart rate, optimally within 50-70/min limits, were chosen due to the minimum impact of such heart rate on QT interval correction formula. QTc data was calculated upon Bazett's formula. QTV and QTVi were calculated upon Berger's formula.

After getting all results they were checked against the following exclusion criteria: 1) revealing that information about patient's chronic illness or drugs therapy was obfuscated, revealing increased fasting serum glucose concentration or ionic disturbances. It was strongly recommended to every patient to visit their GP for further diagnostics, 2) revealing any important deviation in physical examination i.a. blood pressure taken twice at the visit ≥140/ ≥90 mmHg, 3) revealing, upon Holter ECG examination, tachycardia or too numerous artifacts making QT interval assessment incredible, 4) too short total sleep time (< 6 hours) registered on polygraphy.

Out of 187 consecutive patients meeting the inclusion criteria, 66 patients met at least one exclusion criterion, leaving 121 patients for the study analyses.

ELIGIBILITY:
Inclusion Criteria:

* gender: female or male,
* age 35-65 years old,
* visceral obesity,
* lack of acute or chronic diseases that may have an influence on rhythm or conduction disorders,
* not undergoing Continuous Positive Airway Pressure therapy (CPAP) or taking drugs that have or may have an influence on QT interval duration [according to Credible Meds list (Woosley et al, 2019)],
* not consuming grapefruits or grapefruit juice for at least 2 weeks before Holter-ECG examination.

Exclusion Criteria:

* revealing that information about patient's chronic illness or drugs therapy was obfuscated, revealing increased fasting serum glucose concentration or ionic disturbances. It was strongly recommended to every patient to visit their GP for further diagnostics,
* revealing any important deviation in physical examination i.a. blood pressure taken twice at the visit ≥140/ ≥90 mmHg,
* revealing, upon Holter ECG examination, tachycardia or too numerous artifacts making QT interval assessment incredible,
* too short total sleep time (< 6 hours) registered on polygraphy.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out of 187 consecutive patients meeting the inclusion criteria, 66 patients met at least one exclusion criterion, leaving 121 patients for the study analyses.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
A number of patients with visceral obesity and Obstructive Sleep Apnea | one day per each patient
  Polygraphy examination of each patient

SECONDARY OUTCOMES:
A number of patients with visceral obesity and heart rhythm disorders occurrence. | Holter ECG - one day per patient
  Holter-ECG monitoring of each patient
Correlation of Obstructive Sleep Apnea and ECG changes among OSA positive and negative patients | 2016-2019
  statistical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Jarecka-Dobroń, PhD, Principal Investigator — NowodworskieMD

IPD SHARING:
Plan to Share IPD: Yes
For a reasonable request the principal intevstigator will share stastical data of studied group.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: As soon as posible after getting the request.
Access Criteria: All requests will be considered by the main investigator and data will be send to the indicated e-mail.

REFERENCES:
- [Background] Alam I, Lewis MJ, Lewis KE, Stephens JW, Baxter JN. Influence of bariatric surgery on indices of cardiac autonomic control. Auton Neurosci. 2009 Dec 3;151(2):168-73. doi: 10.1016/j.autneu.2009.08.007. Epub 2009 Aug 31. PMID 19720569
- [Background] 2. American Academy of Sleep Medicine. International classification of sleep disorders, 2nd ed. Diagnostic and coding manual. Westchester, Illinois: American Academy of Sleep Medicine 2005. Updated November 2015. Darien, IL: American Academy of Sleep medicine, 2016.
- [Background] Sleep-related breathing disorders in adults: recommendations for syndrome definition and measurement techniques in clinical research. The Report of an American Academy of Sleep Medicine Task Force. Sleep. 1999 Aug 1;22(5):667-89. No abstract available. PMID 10450601
- [Background] Arslan E, Yiginer O, Yavasoglu I, Ozcelik F, Kardesoglu E, Nalbant S. Effect of uncomplicated obesity on QT interval in young men. Pol Arch Med Wewn. 2010 Jun;120(6):209-13. PMID 20567204
- [Background] Barta K, Szabo Z, Kun C, Munkacsy C, Bene O, Magyar MT, Csiba L, Lorincz I. The effect of sleep apnea on QT interval, QT dispersion, and arrhythmias. Clin Cardiol. 2010 Jun;33(6):E35-9. doi: 10.1002/clc.20619. PMID 20552591
- [Background] Baumert M, Schlaich MP, Nalivaiko E, Lambert E, Sari CI, Kaye DM, Elser MD, Sanders P, Lambert G. Relation between QT interval variability and cardiac sympathetic activity in hypertension. Am J Physiol Heart Circ Physiol. 2011 Apr;300(4):H1412-7. doi: 10.1152/ajpheart.01184.2010. Epub 2011 Jan 21. PMID 21257917
- [Background] Baumert M, Porta A, Vos MA, Malik M, Couderc JP, Laguna P, Piccirillo G, Smith GL, Tereshchenko LG, Volders PG. QT interval variability in body surface ECG: measurement, physiological basis, and clinical value: position statement and consensus guidance endorsed by the European Heart Rhythm Association jointly with the ESC Working Group on Cardiac Cellular Electrophysiology. Europace. 2016 Jun;18(6):925-44. doi: 10.1093/europace/euv405. Epub 2016 Jan 27. PMID 26823389
- [Background] Baumert M, Smith J, Catcheside P, McEvoy RD, Abbott D, Sanders P, Nalivaiko E. Variability of QT interval duration in obstructive sleep apnea: an indicator of disease severity. Sleep. 2008 Jul;31(7):959-66. PMID 18652091
- [Background] Gami AS, Howard DE, Olson EJ, Somers VK. Day-night pattern of sudden death in obstructive sleep apnea. N Engl J Med. 2005 Mar 24;352(12):1206-14. doi: 10.1056/NEJMoa041832. PMID 15788497
- [Background] Gami AS, Olson EJ, Shen WK, Wright RS, Ballman KV, Hodge DO, Herges RM, Howard DE, Somers VK. Obstructive sleep apnea and the risk of sudden cardiac death: a longitudinal study of 10,701 adults. J Am Coll Cardiol. 2013 Aug 13;62(7):610-6. doi: 10.1016/j.jacc.2013.04.080. Epub 2013 Jun 13. PMID 23770166
- [Background] Haigney MC, Zareba W, Gentlesk PJ, Goldstein RE, Illovsky M, McNitt S, Andrews ML, Moss AJ; Multicenter Automatic Defibrillator Implantation Trial II investigators. QT interval variability and spontaneous ventricular tachycardia or fibrillation in the Multicenter Automatic Defibrillator Implantation Trial (MADIT) II patients. J Am Coll Cardiol. 2004 Oct 6;44(7):1481-7. doi: 10.1016/j.jacc.2004.06.063. PMID 15464332
- [Background] Hinterseer M, Beckmann BM, Thomsen MB, Pfeufer A, Dalla Pozza R, Loeff M, Netz H, Steinbeck G, Vos MA, Kaab S. Relation of increased short-term variability of QT interval to congenital long-QT syndrome. Am J Cardiol. 2009 May 1;103(9):1244-8. doi: 10.1016/j.amjcard.2009.01.011. Epub 2009 Mar 18. PMID 19406266
- [Background] 14. Report of a WHO Expert Consultation. Waist circumference and waist-hip ratio. Geneva, 8-11 Dec 2008.
- [Background] Mathieu P, Poirier P, Pibarot P, Lemieux I, Despres JP. Visceral obesity: the link among inflammation, hypertension, and cardiovascular disease. Hypertension. 2009 Apr;53(4):577-84. doi: 10.1161/HYPERTENSIONAHA.108.110320. Epub 2009 Feb 23. No abstract available. PMID 19237685
- [Background] Mehra R, Benjamin EJ, Shahar E, Gottlieb DJ, Nawabit R, Kirchner HL, Sahadevan J, Redline S; Sleep Heart Health Study. Association of nocturnal arrhythmias with sleep-disordered breathing: The Sleep Heart Health Study. Am J Respir Crit Care Med. 2006 Apr 15;173(8):910-6. doi: 10.1164/rccm.200509-1442OC. Epub 2006 Jan 19. PMID 16424443
- [Background] Menon A, Kumar M. Influence of body position on severity of obstructive sleep apnea: a systematic review. ISRN Otolaryngol. 2013 Oct 8;2013:670381. doi: 10.1155/2013/670381. PMID 24223313
- [Background] Murabayashi T, Fetics B, Kass D, Nevo E, Gramatikov B, Berger RD. Beat-to-beat QT interval variability associated with acute myocardial ischemia. J Electrocardiol. 2002 Jan;35(1):19-25. doi: 10.1054/jelc.2002.30250. PMID 11786943
- [Background] Myredal A, Karlsson AK, Johansson M. Elevated temporal lability of myocardial repolarization after coronary artery bypass grafting. J Electrocardiol. 2008 Nov-Dec;41(6):698-702. doi: 10.1016/j.jelectrocard.2008.06.004. Epub 2008 Jul 21. PMID 18640686
- [Background] Myredal A, Gao S, Friberg P, Jensen G, Larsson L, Johansson M. Increased myocardial repolarization lability and reduced cardiac baroreflex sensitivity in individuals with high-normal blood pressure. J Hypertens. 2005 Sep;23(9):1751-6. doi: 10.1097/01.hjh.0000179762.93291.94. PMID 16093922
- [Background] Papaioannou A, Michaloudis D, Fraidakis O, Petrou A, Chaniotaki F, Kanoupakis E, Stamatiou G, Melissas J, Askitopoulou H. Effects of weight loss on QT interval in morbidly obese patients. Obes Surg. 2003 Dec;13(6):869-73. doi: 10.1381/096089203322618687. PMID 14738673
- [Background] Romero-Corral A, Caples SM, Lopez-Jimenez F, Somers VK. Interactions between obesity and obstructive sleep apnea: implications for treatment. Chest. 2010 Mar;137(3):711-9. doi: 10.1378/chest.09-0360. PMID 20202954
- [Background] Sosnowski M, Czyz Z, Tendera M. Time and frequency analysis of beat-to-beat R-T interval variability in patients with ischaemic left ventricular dysfunction providing evidence for non-neural control of ventricular repolarisation. Eur J Heart Fail. 2002 Dec;4(6):737-43. doi: 10.1016/s1388-9842(02)00167-8. PMID 12453544
- [Background] Strack C, Fessman D, Fenk S, Waldmann K, Kempinger S, Loew T, et al. QT prolongation is frequently observed in obesity with and without the metabolic syndrome and can be reversed by long term weight reduction. Eur Heart J 2013 34:4287.
- [Background] Viigimae M, Karai D, Pilt K, Pirn P, Huhtala H, Polo O, Meigas K, Kaik J. QT interval variability index and QT interval duration during different sleep stages in patients with obstructive sleep apnea. Sleep Med. 2017 Sep;37:160-167. doi: 10.1016/j.sleep.2017.06.026. Epub 2017 Jul 22. PMID 28899529
- [Background] Vrtovec B, Starc V, Starc R. Beat-to-beat QT interval variability in coronary patients. J Electrocardiol. 2000 Apr;33(2):119-25. doi: 10.1016/s0022-0736(00)80068-0. PMID 10819405
- [Background] 28. Woosley R.L., Romero K.A., www.Crediblemeds.org, QTdrugs List, [access date 05 May 2019, AZCERT, Inc. 1822 Innovation Park Dr., Oro Valley, AZ 85755.